CLINICAL TRIAL: NCT00771654
Title: Does the Addition of Phentermine Increase Weight Loss in the Obese After Gastric Band Operation?
Brief Title: Phentermine/Gastric Band Weight Loss Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07-08-01A
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2022-04-21 (Actual); Status verified 2012-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Phentermine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Subjects will be randomized to the daily dosing of either oral Phentermine 37.5mg or placebo to commence at their 2 week follow-up appointment following their gastric band procedure
  Interventions: Other: Placebo
- Phentermine (Experimental): Subjects will be randomized to the daily dosing of either oral Phentermine 37.5mg or placebo to commence at their 2 week follow-up appointment following their gastric band procedure
  Interventions: Drug: Phentermine

INTERVENTIONS:
Drug: Phentermine — Subjects will receive Phentermine 37.5mg everyday for one year
  Other Names: Adipex
  Arms: Phentermine
Other: Placebo — daily for one year
  Arms: Placebo

SUMMARY:
This is a prospective, randomized, double-blind controlled trial. The goal is to show whether the administration of daily oral Phentermine will augment patient weight loss and resolve obesity associated comorbidities following gastric band operation.

ELIGIBILITY:
Inclusion Criteria:

* Adult age 18-65
* BMI 35-55
* Approved for gastric band operation

Exclusion Criteria:

* A known allergy to Phentermine
* Take medications for Attention Deficit Disorder (ADD)
* Monoamine oxidase inhibitors (MAOI)for depression
* Selective serotonin reuptake inhibitor (SSRIs)for depression
* History of heart problems (congested heart failure, coronary artery disease,cardiac stents, cardiac arrhythmias
* Hyperthyroidism
* Glaucoma
* Psychosis
* History of drug abuse
* Uncontrolled hypertension (diastolic >85)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Primary outcomes are total weight loss and excess weight | one year

SECONDARY OUTCOMES:
Secondary outcomes is resolution of preoperative comorbidities | one year

CONTACTS AND LOCATIONS:
Overall Officials: Keith Gersin, MD, Principal Investigator — Wake Forest University Health Sciences